CLINICAL TRIAL: NCT06378892
Title: A Multicenter Single-arm Phase II Interventional Study to Evaluate the Activity and Safety of the Combination of Platinum-pemetrexed Based Chemotherapy Plus Lorlatinib in ALK Positive Non-Small Cell Lung Cancer (NSCLC) With Exclusively Extracranial Disease Progression on Lorlatinib.
Brief Title: A Study to Evaluate the Combination of Platinum-pemetrexed Based Chemotherapy Plus Lorlatinib in ALK Positive Non-Small Cell Lung Cancer (NSCLC) With Exclusively Extracranial Disease Progression on Lorlatinib
Acronym: ALK-PPL
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Centro di Riferimento Oncologico - Aviano (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CRO-2023-78
Record Dates: First submitted 2024-04-10; First posted 2024-04-23 (Actual); Last update posted 2024-04-23 (Actual); Status verified 2024-04

CONDITIONS: Non Small Cell Lung Cancer Metastatic; ALK Gene Mutation
MeSH Terms: interventions — lorlatinib

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Lorlatinib (Experimental): Lorlatinib 100mg once daily. Carboplatin AUC 5 or Cisplatin 75 mg/m^2 for an induction phase of four cycles. Pemetrexed 500 mg/m^2 during the maintenance phase.
  Interventions: Drug: Lorlatinib

INTERVENTIONS:
Drug: Lorlatinib — Platinum-pemetrexed based chemotherapy plus Lorlatinib will be administered for an induction phase of four cycles. The choice between Carboplatin or Cisplatin is entrusted to the clinician. Subsequently, patients with response or stability of disease at radiological assessment will start the maintenance phase with pemetrexed-Lorlatinib in 21-day cycles until progression, unacceptable toxicity, death, or withdrawal of consent.

SUMMARY:
This study aims to evaluate the activity and safety of the combination of platinum-pemetrexed based chemotherapy plus Lorlatinib in ALK positive Non-Small Cell Lung Cancer (NSCLC) with exclusively extracranial disease progression on Lorlatinib. Platinum-pemetrexed based chemotherapy plus Lorlatinib will be administered for an induction phase of four cycles. Subsequently, patients with response or stability of disease at radiological assessment will start the maintenance phase with pemetrexed-Lorlatinib in 21-day cycles until progression, unacceptable toxicity, death, or withdrawal of consent.

DETAILED DESCRIPTION:
This is a multicentre, phase II, interventional, prospective, single arm, non-randomised study focused on ALK+ NSCLC with extracranial progression on Lorlatinib.Treatment phase include the period starting from cycle 1 day 1 visit to discontinuation of study therapy and consists of two phases: induction phase and maintenance phase. Platinum-pemetrexed based chemotherapy plus Lorlatinib will be administered for an induction phase of four cycles. Subsequently, patients with response or stability of disease at radiological assessment will start the maintenance phase with pemetrexed-Lorlatinib in 21-day cycles until progression, unacceptable toxicity, death, or withdrawal of consent.

ELIGIBILITY:
Key Inclusion Criteria:

* Histologically or cytologically confirmed diagnosis of stage IV ALK positive NSCLC.
* Patients must be in progression extracranially on Lorlatinib; Lorlatinib may be in first- or further-line, without limitations regarding previously received therapies.
* Age at the time of signing the informed consent at least 18 years.
* Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1.
* Patients must have measurable disease according to RECIST 1.1 by computed tomography (CT) and magnetic resonance imaging (MRI).
* Radiologically confirmed multiple extracranial progression on Lorlatinib without progression in the central nervous system (CNS) defined as absence of CNS metastasis or CNS metastasis stable on Lorlatinib and/or stereotactic brain irradiation (SBRT).
* Adequate organ function (kidney, bone marrow and liver).
* Estimated life expectancy of at least 3 months irrespective of the diagnosis of ALK+ NSCLC.
* For women of childbearing potential and males with partners of childbearing potential: agreement to remain abstinent (refrain from heterosexual intercourse) or use contraceptive methods that result in a failure rate of < 1% per year during the treatment period and for at least 6 months after the last dose of study drugs.

Key Exclusion Criteria:

* Known hypersensitivity reaction to one of the compounds or substances used in this protocol.
* Diagnosis of any secondary malignancy within the last 3 years except for: adequately treated basal cell or squamous cell skin cancer, carcinoma in situ of the cervix, definitively treated nonmetastatic prostate cancer or patients with another primary malignancy who are definitively relapse-free with at least 3 years elapsed since the diagnosis of the other primary malignancy.
* Patients deemed unsuitable by the investigator for treatment of chemo-Lorlatinib combination.
* Presence of toxicities contraindicating the continuation of therapy with Lorlatinib.
* Concomitant use of potent CYP3A4/5 inducers.

Other inclusion/exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2024-03-15 (Actual); Primary Completion 2028-05 (Estimated); Study Completion 2028-05 (Estimated)

PRIMARY OUTCOMES:
Compare Progression Free Survival between patients treated with Pemetrexed (PT)/pem-based chemotherapy plus Lorlatinib after Lorlatinib versus retrospective data of 3,2 months for patients treated with PT/pem-based chemotherapy after Lorlatinib. | Up to 60 months
  PFS defined as the time from study enrollment to the first documented disease progression or death due to any cause, whichever occurs first.

SECONDARY OUTCOMES:
Intracranial Progression Free Survival (PFS) in patients treated with PT/pem-based chemotherapy plus Lorlatinib after Lorlatinib. | Up to 60 months
  Intracranial PFS defined as time from study enrollment until CNS disease progression or death from any cause.
Overall survival (OS) in patients treated with PT/pem-based chemotherapy plus Lorlatinib after Lorlatinib progression | Up to 60 months
  OS is defined as the time from study enrollment until death from any cause.
Describe the safety of PT/pem-based chemotherapy plus Lorlatinib combination | Up to 60 months
  Frequency and severity of adverse events graded according to the CTCAE version 5.0.

CONTACTS AND LOCATIONS:
Locations (9):
- Italy (9):
  - Centro di Riferimento Oncologico (CRO) IRCCS, Aviano
  - Azienda Ospedaliero-Universitaria Careggi Oncologia Medica, Florence
  - Azienda USL Toscana Nord Ovest Oncologia Medica, Ospedale Versilia, Lido di Camaiore
  - Istituto Romagnolo per lo Studio dei Tumori (IRST) "Dino amadori", Meldola
  - Fondazione IRCCS San Gerardo dei Tintori, Monza
  - IOV Istituto Oncologico Veneto IRCCS, Padua
  - Azienda Ospedaliero-Universitaria di Parma, Parma
  - Azienda Ospedaliera di Perugia, Perugia
  - Azienda Sanitaria Universitaria Friuli Centrale (ASU FC), Udine